CLINICAL TRIAL: NCT00968773
Title: Rebound Hernia Repair Device Trial
Brief Title: Rebound Hernia Repair Device Mesh Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Minnesota Medical Development, Inc. (Industry)
Collaborators: University of Kentucky (Other); Ohio State University (Other)
Responsible Party: Steve Nuss Chief Marketing Officer, Minnesota Medical Development, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rebound HRD
Record Dates: First submitted 2009-08-27; First posted 2009-08-31 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2009-09

CONDITIONS: Inguinal Hernia
Keywords: inguinal hernia; mesh; hernia repair device
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The Rebound hernia repair device with no fixation (Experimental): Competent adults who have a unilateral, bilateral inguinal hernia that is primary in nature.
  Interventions: Device: Rebound HRD
- Standard Hernia Mesh using fixation (Active Comparator): Competent adults who have a unilateral or bilateral inguinal hernia that is primary in nature.
  Interventions: Device: Standard hernia mesh (VitaMesh)

INTERVENTIONS:
Device: Rebound HRD — Laparoscopic TEP inguinal hernia repair using the Rebound HRD and no fixation
  Arms: The Rebound hernia repair device with no fixation
Device: Standard hernia mesh (VitaMesh) — Laparoscopic TEP inguinal hernia repair using standard hernia mesh with fixation
  Other Names: VitaMesh
  Arms: Standard Hernia Mesh using fixation

SUMMARY:
This is a post-market study of the Rebound Hernia Repair Device to further establish the safety, efficacy, and utility of the Rebound Hernia Repair Device in a controlled population. The Rebound Hernia Repair Device will be used for its approved indication in comparison to "standard" hernia mesh. Two-way students t-tests, Chi squared analysis and ANOVA will be used to detect differences in variables. The study is sufficiently powered to detect a 25% difference.

The study data will include quality of life assessments, visual analogue scale , SF-36, Carolinas Comfort Scale), recurrence of hernia (technical failure), use of medications (pain) and complications/adverse events.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years of age
* Unilateral or bilateral inguinal hernia (moderate in size), primary in nature

Exclusion Criteria:

* Unable to provide informed consent
* Assessed as ASA 3 or 4
* Renal failure;creatinine greater than 2.0mg percent
* Ascites as determined by clinical suspicion/ultrasound confirmation
* Known pregnancy
* Femoral hernias
* Diabetes requiring injectable insulin
* Prior lower abdominal surgery through lower midline or Pfannenstiel incision
* TAPP approach
* Requiring anticoagulants during surgery
* Participation in another study involving another device or drug
* Emergent procedures for hernia incarceration and strangulation
* Recurrent inguinal hernias

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-03 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Presence of hernia recurrence | 2 years

SECONDARY OUTCOMES:
Pain and discomfort to patients using VAS | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: John S Roth, MD, Principal Investigator — University of Kentucky; Jeffrey W Hazey, MD, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - University of Kentucky Dept. Of Surgery, Lexington, Kentucky
  - The Ohio State Medical Center, Dept. of Surgery, Columbus, Ohio